CLINICAL TRIAL: NCT04412590
Title: Pilot Study of the Vermont Family Based Approach in Primary Care Pediatrics at the University of Vermont Medical Center
Brief Title: Pilot Study of the Vermont Family Based Approach in Primary Care Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, James Hudziak, Professor of Psychiatry, Medicine, Pediatrics, and Communication Sciences & Disorders; Director of the Vermont Center for Children, Youth & Families, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHRMS 16-004
Record Dates: First submitted 2015-09-09; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Psychiatric Disorder
Keywords: Health Promotion; Prevention; Mental health; Quality of life; Pediatrics; Wellness; Preventive Medicine; Preventive Psychiatry; Patient Participation; Health Literacy; Patient Activation; Patient Engagement; Emotional Health; Behavioral Health
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being; Patient Participation | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vermont Family Based Approach (Experimental): The VFBA group was offered a variety of supports and services to help them achieve and maintain wellness and address emotional behavioral challenges.
  All families partnered with a Family Wellness Coach (FWC) to design and implement a comprehensive program of family health and wellness with an emphasis on nutrition, exercise, music training, mindfulness, decreasing screen time, and positive parenting.
  Families with a child or parent experiencing significant emotional and behavioral problems were also partnered with Focused Family Coaches (FFCs) and Family Based Psychiatrists (FBPs). FFCs and FBPs respectively provided evidence-based psychotherapy and psychiatric care from the family perspective.
  Families also were also offered health promotion programs, including music lessons for all family members, behavioral parent training, yoga and mindfulness training, and nutrition coaching.
  Interventions: Other: Vermont Family Based Approach
- Control (Active Comparator): The Control Group received pediatric care as usual.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: Vermont Family Based Approach — Comprehensive and individualized program to promote emotional health and wellbeing in families using evidence-based health promotion, prevention and intervention.
  Other Names: VFBA
  Arms: Vermont Family Based Approach
Other: Treatment as Usual — Pediatric care as usual.
  Other Names: TAU
  Arms: Control

SUMMARY:
This pilot randomized controlled trial of the Vermont Family Based Approach (VFBA) tested the feasibility of the VFBA in primary care pediatrics and its effects on children's and parents' emotional and behavioral problems and health-related quality of life. The VFBA is a public health framework for evidence-based health promotion, prevention, and treatment that is delivered from the family perspective and emphasizes emotional and behavioral health. The VFBA group received the VFBA intervention, while the Control group received pediatric primary care as usual.

DETAILED DESCRIPTION:
To enhance the health of our communities, we need approaches to healthcare delivery that focus on the entire family, recognize the central role of emotional and behavioral health in relation to all health, use evidence-based health promotion in addition to evidence based treatment of existing problems, and intervene early in children's life.

The VFBA is a public health framework for evidence-based health promotion, prevention, and treatment that is delivered from the family perspective and emphasizes emotional and behavioral health.

The study was a pilot RCT of the VFBA in a primary care pediatrics clinic. The goals of the study were to test whether the VFBA would (1) be feasible in primary care pediatrics and (2) would lead to improved emotional and behavioral health and health-related quality of life or children and parents. Families were recruited at the pediatric clinic and randomized to the VFBA or Control conditions.

The VFBA group received family-based assessment of emotional and behavioral health and family functioning, family wellness coaching, and a menu of cost-free wellness activities, such as parent and child violin instruction, yoga and mindfulness training, and nutrition counseling. Where indicated by results of family-based assessment, families in the VFBA group also received family-based, evidence-based psychotherapy and psychiatric care. Families in the Control group received pediatric primary care, as usual.

ELIGIBILITY:
Inclusion Criteria:

* Families with a 3 - 15 year-old child who receives his/her primary care at the University of Vermont Pediatric Primary Care Clinic

Exclusion Criteria:

* Families with a target child in the legal custody of the State of Vermont
* Families where the parents' proficiency in English is not sufficient to participate in the protocol without an interpreter

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility Index 1 | during study enrollment
  descriptive statistics for the number of family visits with FWCs
Feasibility Index 2 | during study enrollment
  descriptive statistics for the number of family visits with FFCs
Feasibility Index 3 | during study enrollment
  number of health and wellness supports and services the family engaged with

SECONDARY OUTCOMES:
Children's Emotional and Behavioral Problems | Baseline, 12 month assessment (final assessment)
  The Child Behavior Checklist (CBCL) Total Problems Score (Range: 0-224; higher scores indicate more emotional and behavioral problems)
Children's Health Related Quality of Life | Baseline, 12 month assessment (final assessment)
  The Child Health Questionnaire for Parents - Short Form (CHQ-SF) General Health Perceptions (Range: 0-100; higher scores indicate greater health-related quality of life)
Parents' Emotional and Behavioral Problems | Baseline, 12 month assessment (final assessment)
  The Adult Self-Report (ASR) Total Problems Score (Range: 0-224; higher scores indicate higher levels of emotional and behavioral problems)
Health Related Quality of Life of Caregivers | Baseline, 12 month assessment (final assessment)
  The MOS 36-item Short-Form Health Survey (MOS-36) General Health Scale (Range: 0-100; higher scores indicate higher health-related quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: James J Hudziak, MD, Principal Investigator — University of Vermont Medical Center
Locations (1):
- Vermont Center for Children, Youth & Families, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Achenbach, T. M., & Rescorla, L. A. (2003). Manual for the ASEBA Adult Forms & Profiles. Burlington, VT: University of Vermont, Research Center for Children, Youth, & Families.
- [Background] Achenbach, T.M., & Rescorla, L.A. (2003). Manual for the ASEBA School-Age Forms & Profiles. Burlington, VT: University of Vermont, Research Center for Children, Youth & Families.
- [Background] Achenbach, T.M., & Rescorla, L.A. (2000). Manual for the ASEBA Preschool Forms & Profiles. Burlington, VT: University of Vermont, Research Center for Children, Youth, and Families.
- [Background] Christensen P. The health-promoting family: a conceptual framework for future research. Soc Sci Med. 2004 Jul;59(2):377-87. doi: 10.1016/j.socscimed.2003.10.021. PMID 15110427
- [Background] Hudziak, J.J., & Bartels, M. (2008). Genetic and environmental influences on wellness, resilience, and psychopathology: A family-based approach for promotion, prevention, and intervention. In J.J. Hudziak (Ed.), Developmental psychopathology and wellness: Genetic and environmental influences. (pp. 267-286). New York, NY: American Psychopathological Association.
- [Background] McHorney CA, Ware JE Jr, Raczek AE. The MOS 36-Item Short-Form Health Survey (SF-36): II. Psychometric and clinical tests of validity in measuring physical and mental health constructs. Med Care. 1993 Mar;31(3):247-63. doi: 10.1097/00005650-199303000-00006. PMID 8450681
- [Background] McHorney CA, Ware JE Jr, Lu JF, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. Med Care. 1994 Jan;32(1):40-66. doi: 10.1097/00005650-199401000-00004. PMID 8277801
- [Background] Raat H, Botterweck AM, Landgraf JM, Hoogeveen WC, Essink-Bot ML. Reliability and validity of the short form of the child health questionnaire for parents (CHQ-PF28) in large random school based and general population samples. J Epidemiol Community Health. 2005 Jan;59(1):75-82. doi: 10.1136/jech.2003.012914. PMID 15598731
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Hudziak J, Ivanova MY. The Vermont Family Based Approach: Family Based Health Promotion, Illness Prevention, and Intervention. Child Adolesc Psychiatr Clin N Am. 2016 Apr;25(2):167-78. doi: 10.1016/j.chc.2015.11.002. Epub 2016 Jan 19. PMID 26980122